CLINICAL TRIAL: NCT01730014
Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneous NNC0148-0000-0287 in Healthy Subjects and in Subjects With Type 1 Diabetes
Brief Title: A Trial Investigating the Safety, Tolerability, and Distribution and Activity in the Body of NNC0148-0000-0287 Injected Under the Skin in Healthy Subjects and in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN1436-3955; 2011-005172-41 (EudraCT Number); U1111-1125-2924 (Other: WHO)
Record Dates: First submitted 2012-11-06; First posted 2012-11-21 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Glargine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Trial part 1 (Experimental)
  Interventions: Drug: 148-0287-A-4.2mM-cartridge; Drug: placebo
- Trial part 2, treatment A (Experimental)
  Interventions: Drug: 148-0287-A-4.2mM-cartridge; Drug: sodium chloride 0.9% w/v
- Trial part 2, treatment B (Experimental)
  Interventions: Drug: placebo; Drug: insulin glargine

INTERVENTIONS:
Drug: 148-0287-A-4.2mM-cartridge — In a dose-escalating design, healthy subjects will receive a single dose, injected subcutaneously.
  Arms: Trial part 1
Drug: placebo — In a dose-escalating design, healthy subjects will receive 148-0287-A-placebo-cartridge, injected subcutaneously.
  Arms: Trial part 1
Drug: 148-0287-A-4.2mM-cartridge — In a dose-escalating design, subjects with type 1 diabetes will receive a single dose, injected subcutaneously. Subjects will only be randomised to receive either treatment A or B.
  Arms: Trial part 2, treatment A
Drug: placebo — In a dose-escalating design, subjects with type 1 diabetes will receive 148-0287-A-placebo-cartridge in a single dose, injected subcutaneously. Subjects will only be randomised to receive either treatment A or B.
  Arms: Trial part 2, treatment B
Drug: insulin glargine — In a dose-escalating design, subjects with type 1 diabetes will receive insulin glargine once daily, injected subcutaneously. Subjects will only be randomised to receive either treatment A or B.
  Arms: Trial part 2, treatment B
Drug: sodium chloride 0.9% w/v — In a dose-escalating design, subjects with type 1 diabetes will receive sodium chloride 0.9% w/v, injected subcutaneously daily. Subjects will only be randomised to receive either treatment A or B.
  Arms: Trial part 2, treatment A

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate safety, tolerability, pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of subcutaneous NNC0148-0000-0287 (insulin 287) in healthy subjects and in subjects with type 1 diabetes

ELIGIBILITY:
Inclusion Criteria:

* TRIAL PART 1 (HEALTHY SUBJECTS):
* Healthy male subject
* Age 18-55 years (both inclusive)
* Body mass index 18.0-28.0 kg/m^2 (both inclusive)
* TRIAL PART 2 (SUBJECTS WITH TYPE 1 DIABETES):
* Healthy male subject (with the exception of conditions associated with diabetes mellitus)
* Age 18-64 years (both inclusive)
* Body mass index 18.0-28.0 kg/m^2 (both incl.)
* Type 1 diabetes mellitus (as diagnosed clinically) and treated with multiple daily insulin injections more than 12 months
* HbA1C (glycosylated haemoglobin) below or equal to 8.5 %
* Current daily basal insulin requirement above or equal to 0.2 to below or equal to 0.8 (I)U/kg/day and current total daily insulin treatment below 1.2 (I)U/kg/day
* Fasting C-peptide below 0.3 nmol/L

Exclusion Criteria:

* The receipt of any investigational medicinal product within the last 3 months prior to the start of this trial (screening)
* Significant blood loss (due to donation, surgery or trauma) of more than 500 mL within 3 months prior to the start of this trial (screening) or participating in any other trial involving blood sampling within the last 2 months before the start of this trial (screening)
* Use of any prescription (see specification below for Trial Part 2) or non-prescription medication, including herbal products and non-routine vitamins, within the last 2 weeks before the start of the trial (screening) that will interfere with the pharmacokinetics of insulin 287, as judged by the investigator in agreement with the sponsor. Routine vitamins and occasional use judged by the investigator in agreement with the sponsor. Routine vitamins and occasional use of paracetamol is permitted up to 48 hours prior to dosing
* History of alcoholism or drug abuse (within the last 2 years), or positive result of alcohol or drug screening test
* Currently smoke more than 1 cigarette per day (or the equivalent for other tobacco products) or smoking 1 cigarette or less per day and not considering being able to refrain from smoking or refrain from use of other types of nicotine products (e.g. such as chewing tobacco, nicotine gums) during the in-house periods
* Habitual excessive consumption of methylxanthine-containing (theophylline, caffeine or theobromine) beverages and foods (coffee, tea, soft drinks such as red bull, cola, chocolate) as judged by the investigator
* Excessive consumption of a diet deviating from a normal diet as judged by the investigator
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation in the trial
* Vulnerable subjects (e.g. persons kept in detention)
* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the trial
* ADDITIONAL KEY EXCLUSION CRITERIA TRIAL PART 2 (subjects with type 1 diabetes):
* Current treatment with statins, systemic (oral, intravenous or inhaled) corticosteroids, monoamine oxidase (MAO) inhibitors, non-selective beta-blockers, thyroid hormones, growth hormone and other drugs, which may interfere with glucose metabolism
* Increased risk of thrombosis, e.g. subjects with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the investigator
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event during the last 12 months) or hypoglycaemic unawareness as judged by the Investigator or hospitalisation for diabetic ketoacidosis during the past 6 months before start of this trial (screening)
* Cardiac problems defined as: decompensated heart failure (New York Heart Association (NYHA) class III and IV) at any time, or acute myocardial infarction at any time, or angina pectoris within the last 12 months before start of this trial (screening)
* Proliferative retinopathy or maculopathy and/or severe neuropathy, in particular autonomic neuropathy, as judged by the investigator

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) | From trial product administration until completion of the post-treatment follow-up visit at Day 37

SECONDARY OUTCOMES:
Incidence of hypoglycaemic episodes | From trial product administration until completion of the post-treatment follow-up visit at Day 37
AUC, the area under the serum insulin 287 concentration-time curve | From dosing visit to infinity calculated from a 0-36 days NNC0148-0287 serum concentration-time-curve based on 43 sampling time points
Cmax, the maximum serum insulin 287 concentration | Observed (within 0-36 days)
tmax, the time for maximum serum insulin 287 concentration | Within 0-36 days
Average morning fasting blood glucose (FBG) concentration | From Day 2 to Day 8
Average morning fasting serum C-peptide concentration | From Day 2 to Day 8
Average morning fasting serum free fatty acid (FFA) concentration | From Day 2 to Day 8
Area under the glucose infusion rate (GIR)-time curve | At Day 1-2, 4-5, or 7-8
The maximal GIR (glucose infusion rate) observed | At Day 1-2, 4-5, or 7-8

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com